CLINICAL TRIAL: NCT04136587
Title: The Bacterial Secretome in Crohn's Disease and Ulcerative Colitis
Brief Title: The Bacterial Secretome in IBD
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 17-199 ex 05/06
Record Dates: First submitted 2019-05-10; First posted 2019-10-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colonic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Healthy Controls: Inclusion criteria:
  * Colonoscopy performed for the following indications: anemia, blood in stool, constipation, change in bowel habits, screening for colon cancer, follow up after polyps, weight loss
  * Macroscopic normal colonoscopy except for diverticulosis (without any signs of inflammation), ≤ 3 polyps (except hyperplastic polyps of the colon and rectum), angiodysplasia
  Exclusion criteria:
  * Diagnosis of IBD or any other inflammatory condition of the small and large intestine
  * Diagnosis of irritable bowel syndrome (IBS)
  * Autoimmune disorders
  * Obesity (BMI> 30)
  * Regular intake of NSAIDs (> 2 tablets/ week), immunosuppressants
  * Intake of antibiotics within the last 3 months
  * Intestinal infection by enteric pathogens
  * Probiotic therapy
  Interventions: Other: Colonic fluid collection during endoscopy for analysis of the bacterial secretome
- Crohn's disease: 2 Subgroups: inactive disease (10 patients) and active disease (10 patients)
  Inclusion criteria:
  * Colonoscopy indicated by routine clinical care
  * Established diagnosis of Crohn´s disease (also if established by the study colonoscopy)
  Exclusion criteria:
  • Intestinal infection by enteric pathogens
  Interventions: Other: Colonic fluid collection during endoscopy for analysis of the bacterial secretome
- Ulcerative Colitis: 2 Subgroups: inactive disease (10 patients) and active disease (10 patients)
  Inclusion criteria:
  * Colonoscopy indicated by routine clinical care
  * Established diagnosis of ulcerative colitis (also if established by the study colonoscopy)
  Exclusion criteria:
  • Intestinal infection by enteric pathogens
  Interventions: Other: Colonic fluid collection during endoscopy for analysis of the bacterial secretome
- Colorectal carcinoma: Inclusion criteria:
  • Diagnosis of a lesion with suspicion for colorectal cancer during endoscopy which is confirmed later by histology
  Exclusion criteria:
  • None
  Interventions: Other: Colonic fluid collection during endoscopy for analysis of the bacterial secretome
- Colitis/Enteritis of other origin: Inclusion criteria:
  * Diagnosis of intestinal inflammation at endoscopy or histology
  * E.g.: Infectious colitis /enteritis; ischemic Colitis; microscopic colitis; graft versus host disease (GVHD); NSAID colitis; Colitis of unknown cause
  Exclusion criteria:
  • None
  Interventions: Other: Colonic fluid collection during endoscopy for analysis of the bacterial secretome

INTERVENTIONS:
Other: Colonic fluid collection during endoscopy for analysis of the bacterial secretome — Colonic content will be collected by suction during routine colonoscopy including the residual fluid in the colon and stool contents and also suction of washing fluid (sterile physiologic H2O solution)

SUMMARY:
Secreted bacterial effectors produced by the intestinal microbiota are in part responsible for the proinflammatory effect of the fecal content in inflammatory bowel disease (IBD) patients.

DETAILED DESCRIPTION:
Fecal colonic content will be collected by suction during routine colonoscopy. From the fecal content different fractions (containing soluble bacterial fractions and membrane bound bacterial fractions) will be processed. These bacterial fractions (also termed as bacterial secretome) will be tested for proinflammatory potential in tissue culture assays including epithelial colonic cell lines and dendritic/monocytic cell lines. The main outcome parameter will be the secretion of proinflammatory cytokines from the tissue culture.

For this purpose the investigators will test different groups of patients including patients with active/inactive Crohn's disease or ulcerative colitis, patients with other inflammatory conditions of the colon, patients with colorectal carcinoma and healthy controls undergoing colonoscopy.

ELIGIBILITY:
Group 1 (healthy controls): n=20

Inclusion criteria:

* Colonoscopy performed for the following indications: anemia, blood in stool, constipation, change in bowel habits, screening for colon cancer, follow up after polyps, weight loss
* Macroscopic normal colonoscopy except for diverticulosis (without any signs of inflammation), ≤ 3 polyps (except hyperplastic polyps of the colon and rectum), angiodysplasia

Exclusion criteria:

* Diagnosis of IBD or any other inflammatory condition of the small and large intestine
* Diagnosis of IBS
* Autoimmune disorders
* Obesity (BMI> 30)
* Regular intake of NSAIDs (> 2 tablets/ week), immunosuppressants
* Intake of antibiotics within the last 3 months
* Intestinal infection by enteric pathogens
* Probiotic therapy

Group 2 (Crohn´s disease; CD): n= 20 (10 active CD; 10 inactive CD)

Inclusion criteria:

* Colonoscopy indicated by routine clinical care
* Established diagnosis of Crohn´s disease (also if established by the study colonoscopy)

Exclusion criteria:

• Intestinal infection by enteric pathogens

Definition of active CD Harvey-Bradshaw Index - HBI ≥ 5 and / or Simple Endoscopic Score for Crohn Disease (SES-CD) ≥ 3

Except SES-CD scores resulting from isolated lesions only located at the ileocolonic anastomosis consistent with a modified Rutgeerts score i2a (these patients are considered as endoscopically non active)

Definition of inactive CD

Harvey-Bradshaw Index (HBI) < 5 and Simple Endoscopic Score for Crohn Disease (SES-CD) < 3

Except SES-CD scores resulting from isolated lesions only located at the ileocolonic anastomosis consistent with a modified Rutgeerts score i2a (these patients are considered as endoscopically non active)

Group 3 (Ulcerative colitis, UC): n= 20 (10 active UC; 10 inactive UC)

Inclusion criteria:

* Colonoscopy indicated by routine clinical care
* Established diagnosis of ulcerative colitis (also if established by the study colonoscopy)

Exclusion criteria:

• Intestinal infection by enteric pathogens

Definition of active UC Total Mayo score ≥ 3 and Endoscopic Mayo subscore ≥ 2

Definition of inactive UC Total Mayo score < 3 and Endoscopic Mayo subscore 0 or 1.

Group 4 (Colorectal cancer): n= 10

Inclusion criteria:

• Diagnosis of a lesion with suspicion for colorectal cancer during endoscopy which is confirmed later by histology

Exclusion criteria:

• None

Group 5 (Colitis/Enteritis of different origin): n= 20

Inclusion criteria:

* Diagnosis of intestinal inflammation at endoscopy or histology
* E.g.: Infectious colitis /enteritis; ischemic Colitis; microscopic colitis; GVHD; NSAID colitis; Colitis of unknown cause

Exclusion criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and active and inactive UC patients
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Concentration of proinflammatory cytokines of bacterial fractions in IBD compared to healthy controls | One day
  Measurement of proinflammatory cytokines (f.e.: IL-8) in epithelial and dendritic tissue culture assays

SECONDARY OUTCOMES:
Concentration of proinflammatory cytokines of bacterial fractions in relation to disease activity | One day
  Measurement of proinflammatory cytokines (f.e.: IL-8) in epithelial and dendritic tissue culture assays
Concentration of proinflammatory cytokines of bacterial fractions in relation to disease type | one day
  Measurement of proinflammatory cytokines (f.e.: IL-8) in epithelial and dendritic tissue culture assays
Concentration of proinflammatory cytokines of bacterial fractions in other colonic diseases | One day
  Measurement of proinflammatory cytokines (f.e.: IL-8) in epithelial and dendritic tissue culture assays

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hoegenauer, Prof, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No